CLINICAL TRIAL: NCT04742413
Title: A 12-Month Observational Prospective Cohort Study to Analyze Cardiometabolic Profile Changes to Switch to Lurasidone in Patients With Schizophrenia. RESPECT Study.
Acronym: RESPECT
Status: Terminated | Type: Observational
Why Stopped: Recruitment was not completed
Sponsor: Angelini Farmacéutica (Industry)
Responsible Party: Sponsor
Other Study IDs: ANG-LUR-2020-01
Record Dates: First submitted 2021-01-22; First posted 2021-02-08 (Actual); Last update posted 2022-09-22 (Actual); Status verified 2022-09

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (2):
- A: Patients who are prescribed to switch to lurasidone (lurasidone cohort)
- B: Patients who are prescribed to switch to any other monotherapy SGA (other SGA cohort)

SUMMARY:
A 12-Month Observational Prospective Multicentre Cohort Study based on existing and newly collected data of schizophrenia patients followed-up for one year in secondary care settings (psychiatric services). Schizophrenia patients will be enrolled in a consecutive manner over a period of 6 month into two cohorts according to their prescribing switching treatment: to lurasidone (cohort A) and to another SGA (cohort B).

DETAILED DESCRIPTION:
Study design A 12-Month observational prospective multicentre cohort study based on existing and newly collected data of schizophrenia patients followed-up for one year in secondary care settings (psychiatric services).

Patients will be selected by the specialist when required to switch the SGA therapy for schizophrenia (index data). Schizophrenia patients will be enrolled in a consecutive manner over a period of 6 month into two cohorts:

* Cohort A: patients who are prescribed to switch to lurasidone (lurasidone cohort)
* Cohort B: patients who are prescribed to switch to any other monotherapy SGA (other SGA cohort) The decision to switch the SGA treatment and prescribe the new treatment is done previously and independent from the decision to enter the patient into the study.

Visit 0 will be performed when the investigator consider necessary to perform the treatment switch and patients give their informed consent to participate in the study. All patients will sign the Informed consent before starting the data collection.

The duration of the study will be 12 months of follow-up after switching (visit 0): month 1 (visit 1), month 3 (visit 2), month 6 (visit 3) and month 12 (visit 4). Moreover, the clinical data of the patients recorded previous the index data will be collected in order to ensure that these patients were on an SGA monotherapy for a minimum of 3 months before switching to maximize potential weight gain and dysmetabolic problems that occurs early during the treatment. Preferably, patients have to be on treatment for a year or more before switching so that they have reached a weight plateau.

ELIGIBILITY:
Inclusion Criteria:

1. Female and male patients ≥ 18 years of age.
2. Patients with schizophrenia based on the Diagnostic of Statistical Manual of Mental Disorders, Fifth Edition (DSM-5).
3. Patients currently treated with oral SGA monotherapy for a minimum of 3 months that are prescribed* to switch to another oral SGA medication. Patients will be included in a cohort depending on the switching treatment prescribed:

   * Cohort A: patients who are prescribed to switch to lurasidone (lurasidone cohort)
   * Cohort B: patients who are prescribed to switch to any other monotherapy SGA (other SGA cohort) *Treatment switch and overlap period will be performed according to clinical practice and medical criteria.
4. Written informed consent prior to participation.

Exclusion Criteria:

1. Patients with a known cardiovascular disease or suspected of having a heart disease.
2. Pregnant or breastfeeding women.
3. Patients diagnosed with at least one of the following: depression with psychotic symptoms, schizoaffective disorder, bipolar disorder or organic brain syndromes; Patients with active suicidal ideation or patients who have habitual and sustained consumption of alcohol and / or other toxic substances are also excluded.
4. Patients who had been treated with a long-acting within the last 6 months, or within last year in case of Trevicta®.
5. Concomitant treatments with antipsychotics for insomnia or anxiety (i.e., low doses of quetiapine, etumine, levomepromazine or similar). Concomitant treatment with sedative substances not considered antipsychotics (i.e., benzodiazepines or similar) when they are being taking regularly and at unchanged low doses are allowed.
6. Patients with history of seizures, stroke, neuroleptic malignant syndrome or epilepsy are excluded.
7. Current participation in any clinical trial.
8. Patients for whom further follow-up is not possible at the enrolling site.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients ≥ 18 years old, with schizophrenia based on the DSM-5, treated with oral SGA monotherapy for a minimum of 3 months before switching to lurasidone or another SGA, will be included.
Sampling Method: Probability Sample
Enrollment: 9 (Actual)
Dates: Start 2020-12-29 (Actual); Primary Completion 2022-02-15 (Actual); Study Completion 2022-03-15 (Actual)

PRIMARY OUTCOMES:
To analyze cardiometabolic profile changes based on metabolic syndrome factors changes from baseline to visit 2. | Month 3
  Body mass index, BMI (kg/m^2)
To analyze cardiometabolic profile changes based on metabolic syndrome factors changes from baseline to visit 2. | Month 3
  Abdominal perimeter (cm)
To analyze cardiometabolic profile changes based on metabolic syndrome factors changes from baseline to visit 2. | Month 3
  Triglycerides(mg/dL)
To analyze cardiometabolic profile changes based on metabolic syndrome factors changes from baseline to visit 2. | Month 3
  High density lipoproteins-cholesterol (mg/dL)
To analyze cardiometabolic profile changes based on metabolic syndrome factors changes from baseline to visit 2. | Month 3
  systolic blood pressure (mm Hg)
To analyze cardiometabolic profile changes based on metabolic syndrome factors changes from baseline to visit 2. | Month 3
  Diastolic blood pressure (mm Hg)
To analyze cardiometabolic profile changes based on metabolic syndrome factors changes from baseline to visit 2. | Month 3
  fasting glucose levels (mg/dL)

SECONDARY OUTCOMES:
To evaluate effectiveness from baseline. | Month 3, month 6 and month 12
  To evaluate effectiveness based on Brief Psychiatric Rating Scale scores from baseline. Smaller scores mean a better outcome. Min: 24; Max:168
To evaluate effectiveness from baseline. | Month 3, month 6 and month 12
  To evaluate effectiveness based on Clinical Global Impressions Ratings scores from baseline. Smaller scores mean a better outcome
Analyze cardiometabolic profile changes based on metabolic syndrome factors | Month 3, month 6 and month 12
  Body Mass Indez (kg/m^2) changes from baseline to visit 1, 3 and 4.
Analyze cardiometabolic profile changes based on metabolic syndrome factors | Month 3, month 6 and month 12
  abdominal perimeter (cm) changes from baseline to visit 1, 3 and 4.
Analyze cardiometabolic profile changes based on metabolic syndrome factors | Month 3, month 6 and month 12
  Triglycerides (mg/dL) changes from baseline to visit 1, 3 and 4.
Analyze cardiometabolic profile changes based on metabolic syndrome factors | Month 3, month 6 and month 12
  High Densitity Lipoproteins - cholesterol (mg/dL) changes from baseline to visit 1, 3 and 4.
Analyze cardiometabolic profile changes based on metabolic syndrome factors | Month 3, month 6 and month 12
  Systolic Blood Preassure (mm Hg) changes from baseline to visit 1, 3 and 4.
Analyze cardiometabolic profile changes based on metabolic syndrome factors | Month 3, month 6 and month 12
  Diastolic Blood Preassure (mm Hg) changes from baseline to visit 1, 3 and 4.
Analyze cardiometabolic profile changes based on metabolic syndrome factors | Month 3, month 6 and month 12
  fasting glucose levels (mg/dL) changes from baseline to visit 1, 3 and 4.
Analyze cardiometabolic profile based on other cardiovascular risk factors | Month 1, month 3, month 6 and month 12
  To analyze cardiometabolic profile based on other cardiovascular risk factors (LDL-c (mg/dL), TC (mg/dL), HbA1c (%), creatinine (mg/dL), eGFR and prolactin (ng/ml) changes from baseline
Analyze cardiometabolic profile based on other cardiovascular risk factors | Month 1, month 3, month 6 and month 12
  Low Density Lipoproteins - cholesterol (mg/dL) changes from baseline
Analyze cardiometabolic profile based on other cardiovascular risk factors | Month 1, month 3, month 6 and month 12
  Total Cholesterol (mg/dL) changes from baseline
Analyze cardiometabolic profile based on other cardiovascular risk factors | Month 1, month 3, month 6 and month 12
  Hemoglobin A1c protein (%) changes from baseline
Analyze cardiometabolic profile based on other cardiovascular risk factors | Month 1, month 3, month 6 and month 12
  creatinine (mg/dL) changes from baseline
Analyze cardiometabolic profile based on other cardiovascular risk factors | Month 1, month 3, month 6 and month 12
  prolactine (ng/mL) changes from baseline
QTc levels | Month 12
  To compare QTc levels from baseline to visit 4 (month 12)
Change in weight | Month 1, month 3, month 6 and month 12
  To analyze the percentage of change in weight (kg) from baseline.
Health-related quality of life (HRQoL) changes based on patient reported outcomes | Month 3, month 6 and month 12
  To describe the health-related quality of life (HRQoL) changes based on patient reported outcomes from baseline.
Health resources use | Month 3, month 6 and month 12
  To analyze the health resources use during the study.
Evaluate safety and tolerability | through study completion, an average of 1 year
  To evaluate safety and tolerability based on adverse events / adverse drug reactions (serious and non-serious) reported along the study
Reason for SGA discontinuation | through study completion, an average of 1 year
  To evaluate the reason for SGA discontinuation by antipsychotic therapy.

CONTACTS AND LOCATIONS:
Locations (10):
- Spain (10):
  - Hospital Regional de Málaga, Málaga, Andalusia
  - Hospital Son Llatzer, Palma de Mallorca, Balearic Islands
  - Hospital Universitario Son Espases, Palma de Mallorca, Balearic Islands
  - Complejo Asistencial Universitario de León, León, Castille and León
  - H. U. Salamanca, Salamanca, Castille and León
  - Complejo Asistencial de Zamora, Zamora, Castille and León
  - CHU Santiago, Santiago de Compostela, Galicia
  - Hospital Álvaro Cunqueiro, Vigo, Galicia
  - Hospital 12 de Octubre, Madrid
  - Hospital Universitario la Paz, Madrid

IPD SHARING:
Plan to Share IPD: No